CLINICAL TRIAL: NCT04364295
Title: Evaluating Real-World Spine Outcomes for Spinal and Orthobiologics Products From Around the World
Brief Title: Stronger Together Global Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SS-GR-1902
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Implanted with SeaSpine spinal or orthobiologics product: Standard of Care Registry- Patients must have been implanted with at least one SeaSpine product
  Interventions: Device: Spinal Surgery with SeaSpine product

INTERVENTIONS:
Device: Spinal Surgery with SeaSpine product — Implanted with SeaSpine spinal or orthobiologic product

SUMMARY:
A global, prospective, non-randomized, multicenter, observational, post-market, medical record review registry evaluating real-world evidence for SeaSpine products.

DETAILED DESCRIPTION:
To gain observational, prospective, real-world clinical, and radiographic data in order to evaluate continued safety and performance following the implantation of SeaSpine products.

ELIGIBILITY:
Inclusion Criteria:

* Have been treated with at least one SeaSpine product.
* Have obtained radiographic imaging, as part of the standard of care, at the following time points: preoperative and postoperative.
* Have obtained at least one preoperative patient-reported outcome measure, as part of the standard of care.
* Patient is planned, per standard of care, to be assessed with radiographic imaging and consistent patient-reported outcome measure(s) from preoperative through at least two scheduled follow-up visits.

Exclusion Criteria:

* Was not implanted with at least one SeaSpine product during operation
* Any other condition that the Investigator determines is unacceptable for enrollment into this registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 2285 patients who were previously implanted with SeaSpine products
Sampling Method: Non-Probability Sample
Enrollment: 2285 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of product failure | 12 months post-operative
  Product failure is defined as product fracture, loosening, gross migration and/or dissociation.

SECONDARY OUTCOMES:
Incidence of product-related Serious Adverse Events (SAEs) related to the spine, fusion or bone healing, and intraoperative and postoperative unanticipated adverse device effects | Intra-operative to 24 months
  Product-related SAEs related to the spine, fusion, or bone will be collected for this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vizesi, PhD, Study Director — SeaSpine Orthopedics Corporation
Locations (2):
- United States (2):
  - Spine Colorado, Durango, Colorado
  - OrthoNeuro, New Albany, Ohio

IPD SHARING:
Plan to Share IPD: No